CLINICAL TRIAL: NCT02995837
Title: Cerebral Blood Flow and Neurocognition in Children With Obstructive Sleep Apnea
Brief Title: Cerebral Blood Flow and Childhood Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-012750; K01HL130719 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; Cerebral Blood Flow; Neurocognition
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Wakefulness; Sleep

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea Syndrome (OSAS): The study duration is estimated at 12-14 months approximately. However, this will depend on the timing of treatment as they will undergo testing pre- and post-OSAS treatment. Participation will entail a total of 8 visits including:
  Pre-treatment - neurocognitive testing, and CBF during wakefulness testing duration is one full day. The CBF nighttime testing is one full night.
  Post-treatment - Six to twelve weeks after clinically indicated surgical treatment, OSAS participants will have a repeat baseline polysomnogram (one full night) to assess for residual OSA. Six and twelve months after the surgical treatment, the sleep study with the nighttime CBF testing, as well as the daytime neurocognitive testing and CBF testing will be repeated to assess for changes.
  Interventions: Other: Sleep Study; Other: Neurocognitive Testing; Other: CBF During Wakefulness; Other: CBF During Sleep
- Controls: The study will include 7 total visits for controls: a baseline sleep study to ensure normalcy, three full days of neurocognitive testing and CBF testing (baseline, 6 and 12 months), and three sleep studies with CBF testing (baseline, 6 and 12 months). A daytime visit and one night time visit may be scheduled during a 24-hour period if the participant and family wish so. Otherwise, they will be scheduled on separate days.
  Interventions: Other: Sleep Study; Other: Neurocognitive Testing; Other: CBF During Wakefulness; Other: CBF During Sleep

INTERVENTIONS:
Other: Sleep Study — Overnight, video-recorded sleep study will be performed in a dedicated pediatric sleep lab. Sleep architecture, apneas and hypopneas, arterial oxygen saturation and end-tidal carbon dioxide tension will be evaluated during the sleep study. Safety measures including arterial oxygen saturation using pulse oximetry, EEG and EKG will be continuously monitored during the study.
  Other Names: Polysomnography
Other: Neurocognitive Testing — Cognitive and behavioral measures including intelligence, attention, working memory, and processing speed will be assessed by a trained psychologist.
Other: CBF During Wakefulness — Cerebral blood flow (CBF) will be measure using Diffuse optical and correlation spectroscopy (DOS/DCS), a non-significant risk device used to collect data for this study but not being tested as part of the protocol. Light sources and detectors which are embedded in a rubber pad will be attached to the subject's head in order to record right and left hemispheric cerebral blood flow, total hemoglobin concentration and tissue oxygen saturation. Measurements will be continuously recorded during the study and averaged for purposes of statistical analysis. With DOS/DCS in place, ventilatory response to hypercapnia will be determined using the rebreathing technique, a standard clinical test. While CBF is being measured, subjects will wear nose clips and sit comfortably breathing through a mouthpiece while the level of carbon dioxide is adjusted over a 3-4 minute period. Oxygen and carbon dioxide levels will be carefully monitored throughout the testing.
  Other Names: Cerebral Blood Flow Testing During Hypercapneic Ventilatory Response (Daytime/Wakefulness)
Other: CBF During Sleep — This is the same as the CBF testing during wakefulness/daytime except that it will be done during a sleep study performed with a continuous positive airway pressure (CPAP) mask not nose clips and a mouthpiece. With DOS/DCS in place, ventilatory response to hypercapnia will be determined using the rebreathing technique. While CBF is being measured, OSAS subjects will receive an individualized positive pressure aimed at treating obstructive sleep apnea and controls will receive a standard pressure. End-tidal carbon dioxide will be measured via a port in the mask. A constant flow of carbon dioxide will be introduced to the circuit, a slowly adjusted until the patient arouses or for a maximum of 3 minutes, whichever occurs first. One trial will be attempted in each sleep stage (slow-wave sleep and rapid-eye-movement) with a minimum of 15 minute of breathing room air between challenges. Oxygen and carbon dioxide levels will be carefully monitored throughout the testing.
  Other Names: Cerebral Blood Flow Testing During Hypercapneic Ventilatory Response (Nighttime/Sleep)

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) causes hypoxemia and hypercapnia, which may impair cerebral blood flow and cause deficits in behavior. This is a case-control study designed to investigate cerebral blood flow and neurocognitive function in children with OSAS when compared to these findings from normal children. The study hypothesis is that children with OSAS have an impaired cerebral blood flow during wakefulness and sleep compared to normal controls, and that the degree of this impairment correlates with neurocognitive function.

DETAILED DESCRIPTION:
OSAS is characterized by repetitive occlusion of the upper airway during sleep that results in hypoxemia, hypercapnia and arousal from sleep. Children with the obstructive sleep apnea syndrome (OSAS) have impaired behavior and cognition compared to normal controls. Previous studies in adults with OSAS have shown significant alterations of cerebral blood flow during wakefulness and sleep and our preliminary data showed blunted cerebral blood flow response to hypercapnia in children with OSAS during wakefulness. However, it is unknown whether children with OSAS also have impaired cerebral blood flow during sleep. It is also unknown whether the deficits in behavior and cognition in children are associated with cerebral blood flow dysregulation.

This study will investigate whether the changes in cerebral blood flow during wakefulness and sleep elicited by hypercapneic challenge, differ in children with OSAS compared to normal controls. Additionally the study will evaluate the changes in cerebral blood flow during wakefulness and sleep elicited by hypercapneic challenge in children with OSAS before and after treatment (adenotonsillectomy, adenoidectomy, or tonsillectomy). Finally, the study will investigate whether the changes in cerebral blood flow elicited by the aforementioned testing correlate with neurocognitive outcomes.

Children with OSAS aged 6-12 years will be recruited following a clinical polysomnogram. Normal age- and gender-matched controls will be recruited from the general community.

The primary interventions of this study for the two groups (OSAS and controls) are: sleep studies, neurocognitive testing, measurement of cerebral blood flow by near-infrared spectroscopy during hypercapnic challenges conducted during wakefulness and sleep. In addition, OSAS subjects will be re-tested after clinical treatment of OSAS to evaluate for resolution of OSAS, and all subjects will be re-tested at two separate time points after baseline to compare changes due to the treatment of OSAS versus those occurring secondary to normal development.

ELIGIBILITY:
Inclusion Criteria (OSAS subjects):

1. Age between 6 years and 12 years. The lower limit criterion was selected to include children who can understand and cooperate with testing. The upper limit criterion was selected to avoid overlap with the adult presentation of OSAS.
2. Absence of neurologic, cardiovascular, pulmonary, or any other chronic illness with the exception of well-controlled asthma
3. No prior surgery on the nose, palate or oropharynx including an adenotonsillectomy
4. No current drug intake that may interfere with testing such as sedatives or stimulants
5. No prior treatment of sleep-disordered breathing
6. Polysomnographic recording criteria: subjects with OSAS must have an obstructive apnea hypopnea index (AHI) ≥ 5/hour and be a candidate for clinically-indicated surgical treatment.
7. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria (OSAS Subjects)

1. Previous adenotonsillectomy
2. Previous use of CPAP
3. Craniofacial anomalies that can interfere with upper airway anatomy (e.g., Treacher-Collins syndrome)
4. Genetic syndromes (e.g., Trisomy 21, Prader-Willi)
5. Attention deficit hyperactivity disorder (ADHD) on medication
6. Developmental delay
7. Non-English speaking participants due to the nature of neurobehavioral testing

Inclusion Criteria (Control subjects)

1. Age between 6 years and 12 years. The lower limit criterion was selected to include children who can understand and cooperate with testing. The upper limit criterion was selected to avoid overlap with the adult presentation of OSAS.
2. Absence of neurologic, cardiovascular, pulmonary, or any other chronic illness with the exception of well-controlled asthma
3. No prior surgery on the nose, palate or oropharynx including an adenotonsillectomy
4. No current drug intake that may interfere with testing such as sedatives or stimulants
5. No prior treatment of sleep-disordered breathing
6. Polysomnographic recording criteria: Normal control subjects must have an AHI ≤ 1.5/hour.
7. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria (Control Subjects)

1. Previous adenotonsillectomy
2. Previous use of CPAP
3. Craniofacial anomalies that can interfere with upper airway anatomy (e.g., Treacher-Collins syndrome)
4. Genetic syndromes (e.g., Trisomy 21, Prader-Willi)
5. ADHD on medication
6. Developmental delay
7. Positive Pediatric Sleep Questionnaire
8. Non-English speaking participants due to the nature of neurobehavioral testing

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with OSAS aged 6-12 years will be recruited following a clinical polysomnogram. Normal age- and gender- matched controls will be recruited from the general community.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio E. Tapia, MD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between October 2016 and February 2020. Participants with obstructive sleep apnea were recruited from the Children's Hospital of Philadelphia Sleep Center.
  Control participants were recruited by means of advertisement.
Pre-assignment Details: Screening phase based on the Adaptive Behavior Assessment System 3 (ABAS 3) and sleep study results resulted in 13 screen failures.
Groups:
- Obstructive Sleep Apnea Syndrome (OSAS): - Typically developing children aged 6-12 years with no history of upper airway surgery or previous treatment of obstructive sleep apnea, with an obstructive apnea hypopnea index equal to or greater than 5 events per hour.
- Controls: - Typically developing children aged 6-12 years with no snoring and no history of previous sleep disordered breathing, and an obstructive apnea hypopnea index ≤1.5/hour.
Period: Overall Study
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls
Started | 19 | 15
Completed | 10 | 7
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (3.4) | 10.3 (3) | 9.81 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 18 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 11 | 26
  White | 1 | 0 | 1
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 14 | 32
Apnea hypopnea index, N/hour [Mean (Standard Deviation); unit: events per hour] — The apnea hypopnea index is the sum of apneas and hypopneas divided by the total hours of sleep during the sleep study night
  events per hour | 16.5 (11.9) | 0.74 (0.44) | 9.6 (11.9)
Body mass index z-score [Mean (Standard Deviation); unit: Z-score] — A Z-score of zero represents the population reference mean. Positive Z-scores represent body mass indices above the mean and negative Z-scores represent body mass indices below the mean. A Z-score equal or greater than2 represents obesity.
  Z-score | 1.87 (1.57) | -0.04 (1.52) | 0.91 (1.96)
Oxyhemoglobin saturation nadir during sleep, % [Mean (Standard Deviation); unit: percentage of oxyhemoglobin] — The measure represents the percentage of hemoglobin that is bound to Oxygen. Greater values are better and lower values are worse.
  percentage of oxyhemoglobin | 83.5 (12) | 91.5 (6) | 86.7 (7.1)
Time with oxyhemoglobin saturation < 90% [Mean (Standard Deviation); unit: % of total sleep time] | 1.1 (1.4) | 0.02 (0.06) | 0.6 (1.2)
Sleep duration [Mean (Standard Deviation); unit: % of total sleep time] — This is the percentage of time that the participant slept during the sleep study night. It is calculated by dividing the sleep time in minutes by the sleep opportunity in minutes and multiplying this result by 100. Greater values are better and lower values are worse.
  % of total sleep time | 84.0 (11.8) | 85.6 (7.3) | 84.7 (10)
Stage N1 [Mean (Standard Deviation); unit: % of total sleep time] | 4.81 (4.62) | 1.31 (3.68) | 4.5 (4.9)
Stage N2 [Mean (Standard Deviation); unit: % of total sleep time] | 46.1 (5.1) | 44.4 (7.9) | 44.4 (6.1)
Stage N3 [Mean (Standard Deviation); unit: % of total sleep time] | 29.05 (9.9) | 31 (5) | 31 (7.6)
Stage Rapid Eye Movement [Mean (Standard Deviation); unit: % of total sleep time] | 18.6 (8.39) | 22.7 (5.17) | 20.3 (5.4)
Sleep arousal [Mean (Standard Deviation); unit: Arousals per hour] — Arousal index represents the total number of arousals divided by hours of sleep. It is widely used in sleep literature.
  Arousals per hour | 13.08 (11.91) | 7.84 (3.28) | 12.9 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebral Blood Flow (CBF) at Baseline Between Obstructive Sleep Apnea Syndrome (OSAS) and Controls
Description: To determine whether children with OSAS have impaired blood flow regulation elicited by hypercapneic challenge compared to normal controls at baseline.
Time Frame: Baseline measurements, up to 24 hours
Population: Percentage of change from baseline of cerebral blood flow during hypercapneic challenge is reported in children with OSAS and controls. Unit is % change from baseline within the groups.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls
Number analyzed (Participants) | 18 | 14
percentage of change from baseline | 184 (56) | 209 (109)

2. Secondary Outcome: Comparison of the Change in CBF From Baseline to Study Completion Between OSAS and Control Subjects
Description: Only children who completed 2 or more repeated measurements were included in the analysis. The change in CBF measurements obtained at baseline when compared at 6 and 12 months after baseline for controls and after adenotonsillectomy for OSAS subjects. The slope of the change in CBF over time is reported: Delta CBF/Delta time, units= percentage over year. Minimum values are -100, maximum values +100, positive values mean better outcome.Cerebral blood flow were measured non-invasively while the child was breathing oxygen mixed with carbon dioxide.
Time Frame: Up to 12 Months
Population: Only children who completed 2 or more repeated measurements were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change per year
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls
Number analyzed (Participants) | 12 | 9
percentage change per year | 0.013 (0.04) | -0.083 (0.17)

3. Other Pre Specified Outcome: Association Between CBF Regulation and Severity of OSAS
Description: Children who completed baseline measurements were included. Correlation coefficients between the obstructive apnea hypopnea index and relative change of cerebral blood flow in children with obstructive sleep apnea and Controls are reported.
  The Correlation Coefficient is calculated by dividing the Covariance of the apnea hypopnea index and CBF by the Standard deviation of the apnea hypopnea index and CBF. Units of the standard deviation of CBF= unit of CBF. So, in the correlation coefficient formula, units get canceled. The correlation coefficient does not have any units and can be positive or negative. In this case positive correlation coefficients signal better regulation of CBF.
Time Frame: Up to 12 months
Population: Correlation coefficients between the obstructive apnea hypopnea index and relative change of cerebral blood flow were calculated
Measure: Number; unit: Correlation coefficients
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls
Number analyzed (Participants) | 18 | 14
Correlation coefficients | -0.0018 | 0.37

4. Other Pre Specified Outcome: Behavior Rating Inventory of Executive Function Global Executive Functioning T-score
Description: Children who completed baseline measurements were included. One child in the obstructive sleep apnea arm did not complete the Behavior Rating Inventory of Executive Function testing.
  Behavior Rating Inventory of Executive Function (global executive functioning T score) is reported between the 2 groups. Because this measures uses a T score, a score of 50 is considered average for the population. The scale is 0-100, with higher scores signaling executive functioning impairment. T-scores of 60-64 are in the mildly elevated range, and scores equal to or exceeding 65 are considered to be significantly elevated. The typical standard deviation (SD) observed is 10.
Time Frame: baseline
Population: Only children who completed the Behavior Rating Inventory of Executive Function testing were included in the analysis
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls
Number analyzed (Participants) | 17 | 13
T score | 56.5 (14.1) | 49.7 (11.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study. Participants were enrolled in the study during 12-14 months unless they were lost of follow up
Description: Definition of adverse event and/or serious adverse event, does not differ from ClinicalTrials.gov definitions.
  Adverse events were collected during visits and the research coordinator called participants on monthly basis inquiring about adverse events.
Arm/Group | Obstructive Sleep Apnea Syndrome (OSAS) | Controls
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/14

LIMITATIONS AND CAVEATS:
Recruitment and retention were affected by the COVID-19 pandemic. For example, many participants refused to come back for follow up testing during the pandemic and the access of normal controls to clinical areas was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT02995837/Prot_SAP_000.pdf